CLINICAL TRIAL: NCT05338645
Title: The Effect of Menopause on the Sexual Functions and Marital Adjustment of the Spouses
Brief Title: Sexual Functions and Marital Adjustment for Spouses in Menopause
Acronym: menopause
Status: Completed | Type: Observational
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Principal Investigator, Hitit University
Other Study IDs: 2017-38
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: This study was conducted as a cross-sectional descriptive study in order to determine the effect of menopause on the SFs and marital adjustment of the spouses.

DETAILED DESCRIPTION:
Objective: This study was conducted as a cross-sectional descriptive study in order to determine the effect of menopause on the SFs and marital adjustment of the spouses.

Materials and Methods: The sample of the study consisted of a total of 254 people, 127 of whom were postmenopausal women and their spouses. The data were collected with The Descriptive Information Form (DIF), The Female Sexual Function Scale (FSFS) and the Arizona Sexual Experiences Scale (ASES), The Marital Adjustment Scale (MAS). T test was used for two-group comparison of parametric data, Mann Whitney U test was used for two-group comparison of non-parametric data, and Kruskal Wallis Test was used for non-parametric data comparison of more than two groups. In addition, the relationship between the mean scores of FSFS, ASES and MAS was evaluated with Spearman's rho Correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* The sample of the study consisted of women aged between 45-65,
* who were aged between 45-65,
* had at least 1 year of menopause,
* had no communication barriers,
* volunteered to participate in the research, -lived in the same house with their spouses, -
* had sexual activity in the last four weeks,
* selected using the simple random sampling method.

Exclusion Criteria:

* have diabetes,
* have hypertension,
* have depression

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of this study, which was planned as a cross-sectional descriptive study, consisted of women who applied to the menopause polyclinic of a university hospital between 08.11.2017 and 29.12.2017. The sample of the study consisted of women aged between 45-65 years. Accordingly, the number of couples to be taken into the sample was determined as 125, and a total of 254 individuals, 127 of whom were menopausal women and their spouses, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Descriptive Information Form (DIF) | 3 mounths
  Descriptive Information Form (DIF) was developed by the researcher according to the literature. This form was applied to 20 women who met the inclusion criteria of the research during the pre-application stage and was rearranged in terms of content and language validity (Bozkurt & Sevil, 2016). This form consists of questions to reveal some characteristics of socio-demographic and marital history such as age, education level, employment status, health insurance, monthly total income, marriage age, duration of marriage, and having children. It was composed of 31 questions in total, including questions to reveal some characteristics of menopause and SFs, such as the status and duration of replacement therapy (HRT), post-menopausal sexual problems, and the status of receiving sexual counseling. During the pre-application stage, DIF was applied to 20 women who met the inclusion criteria and was rearranged in terms of scope and language validity.
Female Sexual Functioning Scale (FSFS) | 3 mounths
  Female Sexual Functioning Scale (FSFS) is a 19-item scale developed by Rosen et al. (2000) to measure SFs in women in the last 4 weeks. The scale was adapted into Turkish by Aygın and Eti (2005). The Cronbach Alpha Coefficient of the scale is 0.75, and the Cronbach Alpha coefficient for the subscales is between 0.89 and 0.98 (Aygın & Aslan, 2005). In the structure of the scale; There are 6 sub-dimensions: desire, arousal, lubrication, orgasm, satisfaction, pain or discomfort. Scoring of the answers is between 1-5 points, and not having sexual intercourse in the last 4 weeks is evaluated as 0 points. The highest score that can be obtained from the scale is 95, and the lowest score is 4. After the subscale means are multiplied by the factor loads, the highest score that can be obtained from the scale is 36 and the lowest score is 2. The cut-off point of the scale is 26.55. Those with a score below 26.55 from the scale are considered to be SDs (Aygın & Aslan, 2005).
Arizona Sexual Experiences Scale-Male Form (ASES) | 3 mounths
  Arizona Sexual Experiences Scale Male Form (ASES) is a 5-item Likert-type scale developed by McGahuey et al. (2000) to evaluate SFs in men. The scale was adapted into Turkish by Atilla Soykan (2002). The Cronbach's Alpha coefficient of the scale was determined as 0.89 (Soykan, 2004). In the structure of the scale; There are 5 sub-dimensions: arousal, arousal, penile hardening, ability to reach orgasm, and satisfaction from orgasm. Each item is scored between 1-6 and the total score varies between 5 and 30. Low scores indicate enhanced sexual function and high scores indicate SD. The cut-off point of the scale is 11. A score of 11 and above is considered as SD.
Marriage Adjustment Scale (MAS) | 3 mounths
  Marriage Adjustment Scale (MAS) is a 15-item Likert-type scale developed by Locke and Wallace (1959) to evaluate marital satisfaction and MA level. It was adapted into Turkish by Tutarel and Kışlak (1999) and the Cronbach's Alpha coefficient was found to be 0.83 for men and 0.84 for women. As the score obtained from the scale increases, MA also increases. Accordingly, the lowest score that can be obtained from the scale is 2, and the highest score is 158. The cut-off point of the scale is 43.5. Those who have a score below 43.5 from the scale are considered to have low MA.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Yıldırım, Principal Investigator — Hitit University
Locations (1):
- Fatma Yıldırım, Çorum, Turkey (Türkiye)